CLINICAL TRIAL: NCT05201755
Title: Continuous Positive Airway Pressure (CPAP) Influence on the Evaluation of Basilica Vein Diameter for Catheter Implantation.
Brief Title: Ultrasound Measurements of Basilica Vein Diameter at Room Air Breathing and at Positive Pressure on Healthy Volunteers
Acronym: PEEPVEIN-2021
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Principal Investigator, Massimiliano Pirrone, Medical Doctor, Anesthesiologist, Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: Not assigned
Record Dates: First submitted 2022-01-09; First posted 2022-01-21 (Actual); Last update posted 2022-08-17 (Actual); Status verified 2022-08

CONDITIONS: Ventilation Therapy; Complications

STUDY DESIGN:
Intervention Model Description: Interventional cross-over study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- A (Other): Investigators will evaluate the diameter of the basilica vein and venous flow-velocity after 5 minutes of breathing at room air. Investigators will collect basic vital parameters (heart rate, blood pressure, pulsoximetry).
  Afterwards, the investigators will administer CPAP through a helmet, with the straps placed under the armpits. After 5 minutes, the investigators will collect again ultrasound data (venous diameter of basilica vein, flow-velocity) and basic vital parameters (heart rate, blood pressure, pulsoximetry).
  Then the CPAP helmet will be tied to the bed and the armpit straps removed. After 5 minutes the investigators will collect ultrasound data and basic vital parameters as in the steps before (venous diameter, flow-velocity, heart rate, blood pressure, pulsoximetry). After this three steps, the protocol ends.
  Interventions: Device: CPAP
- B (Other): Same interventions and measurements as A, in different order (breathing room air, then with a CPAP helmet tied to the bed, then with a CPAP helmet fastened with armpit straps).
  Interventions: Device: CPAP
- C (Other): Same interventions and measurements as A, in different order (breathing with a CPAP fastened with armpit straps, breathing with a CPAP helmet tied to the bed and breathing at room air).
  Interventions: Device: CPAP
- D (Other): Same interventions and measurements as A, in different order (breathing with a CPAP helmet tied to the bed, breathing with a CPAP helmet fastened with armpit straps and breathing at room air).
  Interventions: Device: CPAP

INTERVENTIONS:
Device: CPAP — Application of PEEP (positive end-expiratory pressure) through a CPAP Helmet with a set PEEP of 10 cmH2O. It is a very well tolerated and noninvasive device commonly used for ventilatory support.

SUMMARY:
Peripherally Inserted Central Catheters (PICC) and midline placement requires the catheter size to be one third of the venous diameter, or less. However, measurements during CPAP (Continous Positive Airway Pressure) might overestimate the diameter of veins in patients requiring a PICC line.

The investigators will enroll 28 healthy subjects to measure their basilica vein diameter at atmospheric pressure and at 10 cmH2O of Positive End-Expiratory Pressure (PEEP). PEEP will be applied through a CPAP helmet with the straps placed under the arms or tied to the bed.

The investigators will test the hypothesis that positive airway pressure significantly increases vein diameter. Under this hypothesis, the indication of avoiding catheters larger than one third of the vein diameter should be revised, as venous enlargement during PEEP may lead to the placement of inappropriately large catheters.

DETAILED DESCRIPTION:
After consent, the investigators will enroll 28 participants, randomized with a 1:1:1:1 ratio (sealed envelope) to one of the following groups:

A) Room air -> CPAP (armpit straps) -> CPAP (w/o straps) B) Room air -> CPAP (w/o straps) -> CPAP (armpit straps) C) CPAP (armpit straps) -> CPAP (w/o straps) -> Room air D) CPAP (w/o straps) -> CPAP (armpit straps) - > Room air

The investigators will exclude from the study participants with an ASA score (American Society of Anesthesiology) of 3 or more, subjects with a BMI lower than 20 or with a history of pneumothorax or venous thrombosis. Investigators will enroll adult patients only (age > 18).

The primary endpoint is the evaluation of a clinically significant change in venous diameter in subjects breathing at room air or during positive pressure support.

The investigators decided to deliver CPAP through a CPAP Helmet, as this device is noninvasive, very weill tolerated and widely used at the study hospital. CPAP Helmet are provided with armpit straps. Secondary endpoints are the evaluation of venous flow-velocity changes and the influence of placing the helmet straps under the armpits on venous flow dynamics (venous diameter, flow-velocity).

The study is composed of three steps of 5 minutes each. At each step, the investigators will use ultrasound to measure the diameter of basilica vein and venous flow-velocity at the right mid arm, while recording basic vital signs (heart rate, non-invasive blood pressure, pulsoximetry). The investigators will also gather basic biometric data (age, weight, height, gender). At room air, no intervention is given: after 5 minutes, vital signs are collected and the ultrasound measurements performed (basilica vein diameter, venous blood flow-velocity). At CPAP (armpit straps), the subjects will wear a CPAP helmet and receive 10 cmH2O of PEEP (positive end-expiratory pressure), with the helmet straps placed under the subjects' armpit: after 5 minutes, vital signs are collected and the ultrasound measurements performed (basilica vein diameter, venous blood flow-velocity). At CPAP (w/o straps), the helmet is tied to the subjects' bed: after 5 minutes, vital signs are collected and the ultrasound measurements performed (basilica vein diameter, venous blood flow-velocity).

ELIGIBILITY:
Inclusion Criteria:

* ASA 1 or 2
* BMI > 20

Exclusion Criteria:

* History of pneumothorax
* History of venous thrombosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Venous diameter | 15 minutes
  Changes in diameter of the basilica vein (mm) in subjects breathing at room air or breathing at 10 cmH2O of positive end expiratory pressure

SECONDARY OUTCOMES:
Flow-velocity | 15 min
  Changes in venous flow-velocity of the basilica vein (cm/sec) in subjects breathing at room air or breathing at 10 cmH2O of positive end-expiratory pressure
Venous diameter | 15 min
  Changes in venous diameter (mm) in subjects breathing with a CPAP helmet fastened with the straps under the armpits or with the CPAP helmet tied to the bed instead.
Flow-velocity | 15 min
  Changes in venous flow-velocity (cm/sec) in subjects breathing with a CPAP helmet fastened with the straps under the armpits or with the CPAP helmet tied to the bed instead.

CONTACTS AND LOCATIONS:
Overall Officials: Massimiliano Pirrone, MD, Principal Investigator — Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico
Locations (1):
- IRCCS Fondazione Ca' Granda - Ospedale Policlinico Maggiore, Milan, Italy

IPD SHARING:
Plan to Share IPD: No
No plan